CLINICAL TRIAL: NCT00535821
Title: A Multi-center Randomized Comparison of a Minimally-invasive Cardiovascular Hemodynamic Optimization (MiCHO) Protocol Versus Early Goal-Directed Therapy (EGDT) in the Management of Septic Shock Patients Presenting to the Emergency Department
Brief Title: Minimally-Invasive Cardiovascular Hemodynamic Optimization (MiCHO) Versus Early Goal-Directed Therapy (EGDT) in the Management of Septic Shock
Acronym: MiCHO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollement unavailable technology
Sponsor: Loma Linda University (Other)
Collaborators: University of Massachusetts, Worcester (Other); Wayne State University (Other); VA Loma Linda Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, H. Bryant Nguyen, Medical Doctor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57121
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-05

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: Emergency Department; Hemodynamic Optimization; Esophageal Doppler monitoring; Early Goal-Directed Therapy
MeSH Terms: conditions — Sepsis; Shock, Septic; Emergencies | interventions — Central Venous Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MiCHO (Experimental): A 6-hour resuscitation protocol utilizing the esophageal Doppler monitoring (EDM)
  Interventions: Device: Esophageal Doppler monitoring - CardioQ, Deltex Inc
- EGDT (Active Comparator): A 6-hour resuscitation protocol utilizing CVP/ScvO2
  Interventions: Device: Central line with CVP and continuous ScvO2 monitoring

INTERVENTIONS:
Device: Esophageal Doppler monitoring - CardioQ, Deltex Inc — 6-hour hemodynamic optimization of severe sepsis or septic shock guided by EDM
  Arms: MiCHO
Device: Central line with CVP and continuous ScvO2 monitoring — 6-hour hemodynamic optimization of severe sepsis or septic shock guided by CVP and ScvO2 monitoring
  Arms: EGDT

SUMMARY:
Early intervention in the treatment of septic shock, including early goal-directed therapy (EGDT) in the first 6 hours of disease presentation, has been shown to significantly decrease mortality. However, this approach requires invasive hemodynamic monitoring, thus limiting its widespread application in the emergency department setting. A minimally invasive protocol utilizing esophageal Doppler monitoring (EDM) may be of benefit and practical if it is shown to result in similar outcome as EGDT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years old
* Source of infection
* Two or more of systemic inflammatory response syndrome criteria
* Systolic blood pressure < 90 mmHg after a fluid bolus OR lactate >= 4 mmol/L
* A central line has been placed for CVP/ScvO2 monitoring

Exclusion Criteria:

* Pregnancy
* Acute stroke
* Acute cardiogenic pulmonary edema
* Status asthmaticus
* Unstable cardiac dysrhythmia
* Active hemorrhage
* Acute seizure
* Drug overdose
* Trauma
* Requiring immediate surgery
* Do-not-resuscitate status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Bryant Nguyen, MD, Principal Investigator — Loma Linda University
Locations (4):
- United States (4):
  - Loma Linda University, Loma Linda, California
  - VA Loma Linda Health Care System, Loma Linda, California
  - University of Massachusetts, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan

REFERENCES:
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] McKendry M, McGloin H, Saberi D, Caudwell L, Brady AR, Singer M. Randomised controlled trial assessing the impact of a nurse delivered, flow monitored protocol for optimisation of circulatory status after cardiac surgery. BMJ. 2004 Jul 31;329(7460):258. doi: 10.1136/bmj.38156.767118.7C. Epub 2004 Jul 8. PMID 15242867
- [Background] Chytra I, Pradl R, Bosman R, Pelnar P, Kasal E, Zidkova A. Esophageal Doppler-guided fluid management decreases blood lactate levels in multiple-trauma patients: a randomized controlled trial. Crit Care. 2007;11(1):R24. doi: 10.1186/cc5703. PMID 17313691
- [Background] Gunn SR, Fink MP, Wallace B. Equipment review: the success of early goal-directed therapy for septic shock prompts evaluation of current approaches for monitoring the adequacy of resuscitation. Crit Care. 2005 Aug;9(4):349-59. doi: 10.1186/cc3725. Epub 2005 May 27. PMID 16137384

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MiCHO | EGDT
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MiCHO | EGDT | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.5 (10.5) | 60.7 (1.2) | 69.0 (6.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
SBP < 90 or Lactate >= 4 mmol/L [Number; unit: participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: In-hospital mortality
Time Frame: hospital
Measure: Number; unit: participants
Arm/Group | MiCHO | EGDT
Number analyzed (Participants) | 2 | 3
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | MiCHO | EGDT
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No